CLINICAL TRIAL: NCT01549093
Title: A Randomized, Open Label, Controlled Study About Endostar Continued Pumping or Injecting Into Vein Combining With Gemcitabine-Carboplatin Versus Gemcitabine-Carboplatin Alone to Treat Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Endostar Continued Pumping Into Vein Combining With Gemcitabine-Carboplatin to Treat Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Jianhua Chen, professer, Hunan Province Tumor Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HunanPTH022
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Endostar; Continued Pumping into; Gemcitabine; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Endostar -Continued Pumping into+GC (Experimental): Endostar that is Continued Pumping into vein Combining With Gemcitabine -Carboplatin
  Interventions: Drug: Gemcitabine,Carboplatin,Endostar
- Endostar -injecting into +GC (Active Comparator): Endostar that is injecting into vein with Gemcitabine -Carboplatin
  Interventions: Drug: Gemcitabine(G) Carboplatin(C) Endostar
- GC (Active Comparator): Gemcitabine -Carboplatin
  Interventions: Drug: Gemcitabine(G) Carboplatin(C)

INTERVENTIONS:
Drug: Gemcitabine,Carboplatin,Endostar — Gemcitabine(G):1000mg/m2 iv on d1,8 q3w; Carboplatin(C):AUC 5 iv on d1 q3w; Endostar:7.5 mg/m2 Continued Pumping into vein with saline,Each pump use 48hours and the dosage is 7.5mg/m2*2 ,on day 1 to day 14, discontinuancing for 7 days and 21 days is one cycle,Continued using 2-6cycles.
  Arms: Endostar -Continued Pumping into+GC
Drug: Gemcitabine(G) Carboplatin(C) Endostar — Gemcitabine(G):1000mg/m2 iv on d1,8 q3w; Carboplatin(C):AUC 5 iv on d1 q3w; Endostar:7.5 mg/m2 injecting into vein for 4 hours with saline on day 1 to day 14, discontinuancing for 7 days and 21 days is one cycle.Continued using 2-6cycles
  Arms: Endostar -injecting into +GC
Drug: Gemcitabine(G) Carboplatin(C) — Gemcitabine(G):1000mg/m2 iv on d1,8 q3w; Carboplatin(C):AUC 5 iv on d1 q3w; 21 days is one cycle.Continued using 2-6cycles
  Arms: GC

SUMMARY:
The purpose of this study is to determine whether Endostar with Gemcitabine-Carboplatin are more effective than Gemcitabine-Carboplatin alone in the treatment of Non-Small Cell Lung Cancer (NSCLC),and about Endostar ,Compared with intravenous, Continued vein-pumping maby is a more effective way.

DETAILED DESCRIPTION:
Endostar have anti-tumor activity by against vascular endothelial growth factor for initial treatment. This study was designed to evaluate the safety and efficacy of Endostar Continued vein-pumping Combining with Gemcitabine-Carboplatin (GC)chemotherapy in patients with NSCLC,and seeking for more effective injection.

Methods:

In this randomized, open label, 90 patients are planned to be enrolled at random into 3 arms(1:1:1): Experimental: Endostar -Continued Pumping into+Gemcitabine-Carboplatin(GC),Active Comparator: Endostar -injecting into +Gemcitabine-Carboplatin(GC),Active Comparator: Gemcitabine-Carboplatin(GC),

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed NSCLC;
2. primary treatment,inoperable stage III/IV NSCLC;
3. Age of 18-70years; Gender Not Required;
4. Adequate hematologic, renal, and hepatic function ,Specific index as follows:

   liver function: S-Bilirubin ≤1.5 ULN ; Transaminase≤2 ULN. renal function: S-Creatinine ≤1.2 ULN; blood urea nitrogen ≤1.2 ULN . ULN: upper normal limit. Marrow Hemopoietic Function: WBC≥4.0×10^9/l, ANC≥2.0×10^9/l platelet count ≥100×10^9/l, Hb≥100 g/l;
5. ECOG PS 0-2,Life expectancy ≥ 3 months; endure more than two cycle chemotherapy;
6. The patients have explicit lung tumor lesions and the lesions were measurable; (According to the standard of RECIST1.1, they should have at least one of accurately measurable lesions with the largest diameter ≥ 10mm by spiral CT, MRI);
7. No history of serious drug allergy;
8. Informed consent should be obtained before treatment.

Exclusion Criteria:

1. Symptomatic brain metastases with cognitive disorder,bone metastases with complications;
2. Major organ dysfunction and Serious Heart Disease( congestive heart-failure,incontrollable high-risk arrhythmia,unstable angina, valvular disease, myocardial infarct and Resistant hypertension,);
3. Serious complications and investigator consider it is unsuited enrolling;
4. Pregnant or lactating women;
5. Allergic to research drug;
6. participating in other experimental trials and receive the treatment in four weeks;
7. The position that is for observing curative effect have a radiotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | two years

SECONDARY OUTCOMES:
Overall survival (OS) | two years
Clinical benefit rate (CBR) | two years
The level change of CECs,VEGF,TSP-1,VEGFR,P1GF,MVD in blood. | two years
adverse reaction | two years
Time to progression(TTP) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Chen, master, Principal Investigator — Hunan Province Tumor Hospital
Locations (1):
- HuNan province tumor hospital, Changsha, Hunan, China